CLINICAL TRIAL: NCT02577250
Title: Efficacy and Safety of Repeated Intravenous Subanesthetic Ketamine Infusions Among Veterans With Treatment Resistant Depression Comorbid With Chronic Post-Traumatic Stress Disorder: A Proof-of-concept Study
Brief Title: Ketamine Infusions for PTSD and Treatment-Resistant Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cristina Sophia Albott, MD, MA, Minneapolis Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4555-B
Record Dates: First submitted 2015-10-09; First posted 2015-10-16 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Depressive Disorder, Treatment-Resistant; Stress Disorders, Post-Traumatic
Keywords: ketamine; stress disorders, post-traumatic; stress disorders, traumatic; anxiety disorders; mental disorders; adjuvants, anesthesia; analgesics; anesthetics; anesthetics, dissociative; anesthetics, general; anesthetics, intravenous; excitatory amino acid agents; excitatory amino acid antagonists; hypnotics and sedatives; molecular mechanisms of pharmacological action; neurotransmitter agents; peripheral nervous system agents; pharmacologic actions; physiological effects of drugs; psychotropic drugs; sensory system agents; central nervous system agents; central nervous system depressants; depression; depressive disorder; depressive disorder, treatment-resistant; behavioral symptoms; mood disorders; therapeutic uses
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Anxiety Disorders; Mental Disorders; Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Six ketamine infusions (Experimental): Six infusions of 0.5 mg/kg ketamine hydrochloride solution over 2 weeks.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Six infusions of 0.5 mg/Kg of ketamine hydrochloride solution over 2 weeks.

SUMMARY:
The relationship between depression and trauma is well established. Co-occuring depression and post-traumatic stress disorder (PTSD) are associated with more severe symptoms and lower levels of functioning. Veterans with both depression and PTSD have been shown to be at much higher risk of suicide than individuals with only one of these disorders. Ketamine has been shown to have rapid antidepressant effects and also therapeutic action over PTSD symptoms. The purpose of this study is to see whether ketamine, when given as repeated infusions, can produce quick and sustained improvement in depression and PTSD symptoms for individuals who have not had their symptoms effectively treated by current treatments.

DETAILED DESCRIPTION:
The proposed study is a pilot study designed to determine the efficacy and safety of serial ketamine infusions among veterans with treatment-resistant depression (TRD) as well as chronic post-traumatic stress disorder (PTSD). The investigators hypothesize that six infusions of ketamine will be effective in decreasing severity of depressive symptoms and maintaining response.

Participants will be male/female veterans (18 to 75 years old) of any era or military background who suffer from TRD and chronic PTSD. Potential participants will be recruited from Mental Health clinics and screened for eligibility using a two stage process (phone/chart review, followed by interview). Participants will receive six ketamine infusions on a Monday-Wednesday-Friday schedule over 2 weeks. On the day of infusion, participants will be required to stay at the clinical site for 3 hours after the medication has been given. Follow-up visits will occur at different time points over the course of 2 months after the two week infusion period has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female veterans aged 18 to 75 years.
* Participants must have a telephone in their home and ability to hear telephone conversations.
* Participants must meet current DSM-IV criteria for major depressive disorder (MDD), single or recurrent, without psychotic features
* Participants must meet DSM-5 criteria for current post-traumatic stress disorder (PTSD) and have received a diagnosis of PTSD greater than or equal to 3 months prior to assessment.
* Current major depressive episode resistant to treatment.
* If applicable, current antidepressant dosages including augmenting agents and/or frequency and duration of psychotherapy sessions must remain stable for at least 6 weeks prior to beginning of the study.

Exclusion Criteria:

* Inability to speak English
* Inability or unwillingness to provide written informed consent
* Moderate/severe cognitive impairment .
* Current or lifetime diagnosis of psychosis-related disorder, bipolar I or II disorder, substance-induced mood disorder, or any mood disorder due to a general medical condition.
* Current or lifetime diagnosis of a Cluster B disorder.
* History of moderate or severe traumatic brain injury, Parkinson's disease, dementia of any type, multiple sclerosis, seizures or other CNS related disorders.
* History of comorbid substance disorder within 6 months of screening as assessed using the Mini International Neuropsychiatric Interview (MINI), plus positive urine toxicology screen test during baseline assessments.
* Prior use of ketamine as an antidepressant.
* Clinically unstable medical illness that could compromise the patient's ability to tolerate or likely interfere with the study procedures (e.g., history of or current myocardial ischemia or arrhythmias, congestive heart failure, severe pulmonary, renal, or hepatic disease, uncontrolled hypertension)
* Current or within less than 14 days use of barbiturates or monoamine oxidase inhibitors (MAOI).
* History of antidepressant- or substance-induced hypomania.
* History of first degree relative(s) with an Axis I psychotic disorder.
* For women: pregnancy (confirmed by baseline lab test), the initiation of female hormonal treatments within 3 months of screening, or inability or unwillingness to use a medically accepted contraceptive method for the duration of the study.
* Imminent risk of suicidal/homicidal ideation and/or behavior with intent and/or plan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 24 hours post-infusion
Clinical-Administered PTSD Scale (CAPS) | 2 weeks after the first infusion

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | up to 2 months
PTSD Checklist | 24 hours post-infusion
Clinical-Administered PTSD Scale (CAPS) | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Shiroma, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center; Cristina S Albott, MD,MA, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis Va Health Care System, Minneapolis MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Albott CS, Lim KO, Forbes MK, Erbes C, Tye SJ, Grabowski JG, Thuras P, Batres-Y-Carr TM, Wels J, Shiroma PR. Efficacy, Safety, and Durability of Repeated Ketamine Infusions for Comorbid Posttraumatic Stress Disorder and Treatment-Resistant Depression. J Clin Psychiatry. 2018 May/Jun;79(3):17m11634. doi: 10.4088/JCP.17m11634. PMID 29727073